CLINICAL TRIAL: NCT02092402
Title: Fecal Microbiota Transplantation in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Robert Brummer, MD, PhD, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013/180
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Fecal transplantation; microbiota transplantation; irritable bowel syndrome; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fecal transplantation of own stool (Placebo Comparator): Autologous fecal transplantation (own stool)
  Interventions: Other: Fecal transplantation
- Fecal transplantation (stool from donor) (Experimental): Allogeneic fecal transplantation (from donor)
  Interventions: Other: Fecal transplantation

INTERVENTIONS:
Other: Fecal transplantation

SUMMARY:
The purpose of this study is to investigate the effect of fecal microbiota transplantation (FMT) on the symptoms of irritable bowel syndrome (IBS) patients.

ELIGIBILITY:
Inclusion criteria for patients

1. Signed informed consent
2. Fulfilled Rome III diagnostic criteria for IBS, and frequency of IBS pain or discomfort for at least 2 days a week in the last 12 weeks
3. Age: 18-65 years

Exclusion criteria for patients

1. High proportion of butyrate-producing microbiota in fecal samples
2. Known organic gastrointestinal disease (e.g. IBD)
3. Previous complicated gastrointestinal surgery
4. Non-gastrointestinal malignancy
5. Dementia, severe depression, major psychiatric disorder, or other incapacity for adequate cooperation
6. Females who are pregnant or breast-feeding
7. Severe endometriosis
8. Antimicrobial treatment 4 weeks prior to first screening visit
9. Antimicrobial prophylaxis (eg. acne, urinary tract infection)
10. Regular consumption of probiotic products 4 weeks prior to randomization
11. Recently (within the last 3 months) diagnosed lactose intolerance
12. Celiac disease
13. Abuse of alcohol or drugs
14. Any clinically significant disease/condition which in the investigator's opinion could interfere with the results of the trial

Inclusion criteria for donors

1. Signed informed consent
2. High-butyrate producing microbiota in fecal samples
3. Age: 18-65 years

Exclusion criteria for donors

1. Known organic gastrointestinal disease (e.g. IBD, IBS, chronic diarrhea or constipation)
2. Gastrointestinal malignancy or polyposis
3. History of major gastrointestinal surgery (e.g. gastric bypass)
4. Eosinophilic disorders of the gastrointestinal tract
5. Current communicable disease (e.g. upper respiratory tract infection)
6. Known or high risk of infectious diseases such as HIV, hepatitis A, B or C
7. Non-gastrointestinal malignancy
8. Dementia, severe depression, major psychiatric disorder, or other incapacity for adequate cooperation
9. Comorbidities such as metabolic syndrome, autoimmune diseases, allergies
10. Chronic pain syndromes (eg. chronic fatigue syndrome, fibromyalgia)
11. Severe or morbid obesity
12. Use of immunosuppressive or chemotherapy agents
13. Antimicrobial treatment or prophylaxis within the last 6 months
14. Females who are pregnant or breast-feeding
15. Known clinically significant abnormal laboratory values
16. Participation in high-risk sexual behaviors
17. Abuse of alcohol or drugs
18. Tattoo or body piercing within the last 6 months
19. Travel to areas with endemic diarrhea during the last 3 months
20. Positive stool testing for C. difficile toxin, ova, parasites, Giarda antigen, cryptosporidium antigen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2016-11 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Effect of fecal microbiota transplantation on the symptoms of IBS patients using the IBS version of the gastrointestinal symptom rating scale (GSRS-IBS) | 6 months

SECONDARY OUTCOMES:
Effect of fecal transplantation on IBS patients' visceral perception (Pain scores on the visual analogue scale during barostat procedure) | 2 months
Effect of fecal transplantation on IBS patients' composition of mucosal microbiota (HITChip analysis) | 2 months
Effect of fecal transplantation on IBS patients' composition of fecal microbiota (HITChip analysis) | 6 months
Effect of fecal transplantation on IBS patients' mucosal immune cell composition (lymphocyte fingerprinting using flow cytometry) | 2 months
Effect of fecal microbiota transplantation on the symptoms of IBS patients using the IBS - severity scoring system (IBS-SSS) | 6 months
Effect of fecal microbiota transplantation on the symptoms of IBS patients using the health-related quality of life questionnaire for IBS patients (IBS-QOL) | 6 months
Effect of fecal microbiota transplantation on the symptoms of IBS patients using the hospital and anxiety depression scale (HADS) | 6 months
Effect of fecal microbiota transplantation on the general health of IBS patients using the SF-36 survey | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Brummer, MD, PhD, Principal Investigator — University Hospital Örebro, Department of Gastroenterology and Örebro University, School of Health and Medical Sciences, Faculty of Medicine and Health, Örebro, Sweden
Locations (1):
- University Hospital Örebro, Örebro, Sweden